CLINICAL TRIAL: NCT06425978
Title: The Efficacy of the Use of Cellular Matrix / A-CP-HA Kit (Combination of Autologous Platelet-rich Plasma and Non-cross-linked Hyaluronic Acid) Compared to Local Estrogen Therapy (Blissel, Estriol 50 Micrograms/g Vaginal Gel) in Women With Genitourinary Syndrome of Menopause. A Randomized Controlled Trial, With a Second Blind Observer.
Brief Title: Efficacy of the Use of Cellular Matrix/ A-CP-HA Kit
Acronym: CellularMatrix
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Collaborators: Regen Lab SA (Industry)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSD-CEL-2023-11; 2023-507200-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cellular Matrix / A-CP-HA Kit (Experimental): (a combination of autologous platelet-rich plasma and non-cross-linked hyaluronic acid) is a sterile tube designed for use in the preparation of a mixture of PRP and hyaluronic acid, tube is under vacuum allowing the withdrawal of 6 ml of blood and contains: 2 ml of hyaluronic acid gel (20mg/ml, 40 mg per tube) in phosphate buffer. Not crosslinked, hyaluronic acid is obtained from bacterial fermentation, 3 g of inert cell-selector gel, and 0.6 ml of anticoagulant (sodium citrate 4%). Centrifuged at 1,500 g, 3,000 rpm for 5 min. Platelet recovery of more than 70%, granulocyte depletion of 94.3% and red blood cells of 99.5% are achieved.
  Interventions: Drug: Cellular Matrix / A-CP-HA Kit
- Local estrogen therapy (Active Comparator): Blissel, estriol 50 micrograms/g vaginal gel
  Interventions: Drug: Local estrogen therapy (Blissel, estriol 50 micrograms/g vaginal gel)

INTERVENTIONS:
Drug: Cellular Matrix / A-CP-HA Kit — For infiltration, a prior preparation of the region with anesthetic cream is performed, procaine 25 mg/g + lidocaine 25 mg/g (Emla 5% cream) in the vulvar area and vaginal introitus. Occlusion of the area with plastic film is performed for 20 minutes. After asepsis and antisepsis, infiltration is performed with mesotherapy needles 31G 4mm, using the technique of superficial "point-to-point" mesotherapy microinjections, in the vestibule and the first 3 cm of the posterior wall of the vagina.
  Arms: Cellular Matrix / A-CP-HA Kit
Drug: Local estrogen therapy (Blissel, estriol 50 micrograms/g vaginal gel) — Blissel®, Estriol vaginal gel 50 micrograms/g, daily application for 15-21 days in a row, then two times a week for 24 weeks (6 months). Application instructions will be explained to the patients. The gel should be applied in the vagina using an applicator with the marked dose, the full applicator should be inserted into the vagina and emptied, preferably at night.
  Arms: Local estrogen therapy

SUMMARY:
This study is a randomized, controlled, non-inferiority trial, that will be performed on 192 women on Menopause (absence of menstruation for at least 12 months), with diagnostic of genitourinary syndrome of menopause (SGM) and a vaginal health index <15 points, that are sexually active.

Patients will be randomized 1:1, equal number assigned to each of the two treatment groups, to receive treatment with two dose of Cellular Matrix / A-CP-HA Kit (a combination of autologous platelet-rich plasma and non-cross-linked hyaluronic acid) separated for a month, and control group that will receive the standard treatment for SGM, local estrogen therapy (Blissel, estriol 50 micrograms/g vaginal gel).

Both groups will be follow-up for 3 and 6 month afther treatment, a blind observer will assess the application of the validated scale (VHIS, VHI), and the investigators will do the FSD, symptom record, maturation index, follow-up photography and evaluation of adverse events and treatment compliance and adherence.

DETAILED DESCRIPTION:
This study is a randomized, controlled, non-inferiority trial, with a second blind observer, comparing effectiveness of the use of Cellular Matrix / A-CP-HA Kit (a combination of autologous platelet-rich plasma and non-cross-linked hyaluronic acid) to the standard line of treatment, local estrogen therapy (Blissel, estriol 50 micrograms/g vaginal gel) in women with genitourinary syndrome of menopause (SGM). Duration of the study estimated is 24 months.

A total of 192 menopausal women, with absence of menstruation for at least 12 months, ≤70 years old, that are sexually active and who report symptoms and signs of SGM, with a vaginal health index <15 points. Patients will be excluded if are in treatment with systemic or local hormonal treatment in the last 3 months, Tamoxifen or Aromatase inhibitor treatments. Vulvovaginal pathologies (condyloma, vaginal intraepithelial neoplasia, vaginal carcinoma, lichen sclerosus, lichen planus, history of radiation, history of cervical cancer, other gynecologic cancer, or pelvic radiation, or active genital infection (eg. g., bacterial vaginosis, genital herpes, candida). Contraindication for vaginal estrogen therapy. Women with thrombocytopenia or coagulation disorders, systemic infections, STDs, cancer of any type in recent treatment, connective tissue diseases. Women who have had pelvic surgery within 6 months.

Patients will be randomized 1:1, equal number assigned to each of the two treatment groups, to receive treatment with two dose of Cellular Matrix / A-CP-HA Kit (a combination of autologous platelet-rich plasma and non-cross-linked hyaluronic acid), separated for a month, and control group that will receive the standard treatment for SGM, local estrogen therapy (Blissel, estriol 50 micrograms/g vaginal gel).

Patients will interviewed about their medical history, age of menopause, symptoms related and history of treatments. Evaluation of the Vaginal Health Index (VHIS), Vulvar Health Index (VHI), vaginal pH, and vaginal maturation index (vaginal cytology). The intensity of VVA symptoms (vaginal burning, vaginal itching, vaginal dryness, dyspareunia and dysuria) will be measured using a 5-cm visual analog scale (VAS), and a valuation of Female Sexual Distress (FSD) score. Photographic monitoring during all phases of the procedure. Routine laboratory test serology will requested for both groups (valid up to 3 months).

Both groups will be follow-up for 3 and 6 month afther treatment, a blind observer will assess the application of the validated scale (VHIS, VHI), and the investigators will do the FSD, symptom record, maturation index, follow-up photography and evaluation of adverse events and treatment compliance and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Women ≤70 years old
* Women that are sexually active
* Women who report symptoms and signs of SGM, with a vaginal health index (VHIS - Bachmann score) < 15 points.
* Women who understand the Spanish language
* Willing to participate in the study and sign informed consent.

Exclusion Criteria:

* Systemic or local hormonal treatment in the last 3 months
* Tamoxifen or Aromatase inhibitor treatments
* Vulvovaginal pathologies (condyloma, vaginal intraepithelial neoplasia, vaginal carcinoma, lichen sclerosus, lichen planus, history of radiation, history of cervical cancer, other gynecologic cancer, or pelvic radiation, or active genital infection (eg. g., bacterial vaginosis, genital herpes, candida) Contraindication for vaginal estrogen therapy
* Women with thrombocytopenia or coagulation disorders, systemic infections, STDs, cancer of any type in recent treatment, connective tissue diseases.
* Women who have had pelvic surgery within 6 months.
* Women who are unwilling or unable to give informed consent and/or do not comply with the study requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with improved symptomatology. | at 6 months after treatment
  Improvement is defined as having a higher score than the baseline in the Vaginal Health Index (VHIS)

SECONDARY OUTCOMES:
Healing percentage | at 6 months after treatment
  defined as percentage of patients scoring ≥ 15 in the VHIS
Evolution of Vaginal Health Index | at 3-months and 6-months follow-up
Evolution of Vulvar Health Index | at 3-months and 6-months follow-up
Evolution of vaginal pH | at 3-months and 6-months follow-up
Evolution of Vaginal maturation index (vaginal cytology) | at 3-months and 6-months follow-up
Evolution of intensity of VVA symptoms (vaginal burning, vaginal itching, vaginal dryness, dyspareunia, and dysuria) | at 3-months and 6-months follow-up
  measured using a 5-cm visual analog scale (VAS)
Incidence of adverse events and serious adverse events | at 3-months and 6-months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.dexeus.com